CLINICAL TRIAL: NCT03390257
Title: Safety and Effectiveness Evaluation of the Sinusway™ Device for Endoscopy of the Nasal Cavity and Paranasal Sinuses in Conjunction With Sinus Balloon Dilation
Brief Title: Study to Evaluate the Safety and Initial Effectiveness of the Sinusway™ for Endoscopy of Sinuses in Conjunction With BSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 3NT Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SD001
Record Dates: First submitted 2017-12-20; First posted 2018-01-04 (Actual); Results first posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-10

CONDITIONS: Sinusitis
Keywords: Endoscopy, BSD
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- 3NT flexible endoscope (Experimental): Evaluation of 3NT flexible endoscope in terms of access and evaluation of the nasal anatomy
  Interventions: Device: 3NT flexible endoscope

INTERVENTIONS:
Device: 3NT flexible endoscope — The nasal anatomy will be accessed and viewed with the device during Balloon Sinus Dilation
  Other Names: Balloon sinus dilation

SUMMARY:
3NT flexible endoscope is a single-use disposable handheld endoscope that provides a means to visualize the nasal cavity and paranasal sinus space and deliver irrigation to treat the sinus ostia and spaces within the paranasal sinus cavities for diagnostic and therapeutic procedures

DETAILED DESCRIPTION:
The rationale behind this feasibility study is to show that access and visualization of the nasal anatomy and paranasal sinuses (Maxillary, Frontal and Sphenoid sinuses) in conjunction with Balloon Sinus Dilation in patients suffering from symptoms attributable to sinusitis is feasible in the office and operating room settings; This is an essential step in the development of a combined dilation and visualization system that will allow visualization, dilation and lavage of the sinuses via their natural ostia during an office visit, and minimize radiation exposure, antibiotic use, multiple office visits, and cost.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient indicated for balloon sinus dilation procedure by the ENT specialist
2. Patient age: adult (>18 years old)
3. Patients in general good health in the opinion of the investigator as determined by medical history and physical examination
4. A patient who is able to understand the requirements of the study, is willing to comply with its instructions and schedules, and agrees to sign the informed consent

Exclusion Criteria:

1. Known history of any significant medical disorder, which in the investigator's judgment contraindicates the patient's participation
2. Patients with known current or previous bleeding disorder receiving anticoagulants (e.g., chronic Coumadin treatment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2019-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Johnson, MD, Principal Investigator — SF Otolaryngology
Locations (2):
- United States (2):
  - SF Otolaryngology, San Francisco, California
  - Ogden Clinic, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 3NT Flexible Endoscope
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 3nt Flexible Endoscope
Number analyzed (Participants) | 14
Age, Continuous [Mean (Full Range); unit: years] | 56.6 [21 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Device Effects
Description: Number of Adverse Device Effects is expected to be similar to the number reported in literature for Nasal Endoscopy
Time Frame: 4 hours
Measure: Number; unit: events
Groups:
- 3NT Flexible Endoscope: Evaluation of 3NT flexible endoscope in terms of access and evaluation of the nasal anatomy
  3NT flexible endoscope: The nasal anatomy will be accessed and viewed with the device during Balloon Sinus Dilation
  No Adverse events were reported during this study.
Arm/Group | 3NT Flexible Endoscope
Number analyzed (Participants) | 14
events | 0

2. Secondary Outcome: Percent of Sinuses Accessed and Visualized Successfully
Description: Physician evaluation of the ability to access and visualize the paranasal sinuses. will be recorded as done/not done/failed
Time Frame: 1 hour
Measure: Number; unit: percentage of sinuses
Arm/Group | 3NT Flexible Endoscope
Number analyzed (Participants) | 14
percentage of sinuses
  Maxillary sinus | 60.5
  Frontal sinus | 100
  Sphenoid sinus | 68.5

3. Secondary Outcome: User Satisfaction (1-bad, 5-good)
Description: Physician satisfaction questionnaire
  (1-bad, 5-good)
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: score on a scale 1-5
Arm/Group | 3NT Flexible Endoscope
Number analyzed (Participants) | 14
score on a scale 1-5
  Image quality | 4 (0.39)
  Ease of use | 4.4 (0.5)
  Lavage | 4.5 (0.52)
  Tolerability to patient | 4.6 (1.13)
  Maxillary sinus access | 4.8 (0.44)
  Frontal sinus access | 4.6 (0.52)
  Sphenoid sinus access | 4.7 (0.52)

ADVERSE EVENTS:
Time Frame: day of procedure
Arm/Group | 3NT Flexible Endoscope
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-03): https://cdn.clinicaltrials.gov/large-docs/57/NCT03390257/Prot_001.pdf
  • Informed Consent Form (2017-07-31): https://cdn.clinicaltrials.gov/large-docs/57/NCT03390257/ICF_002.pdf